CLINICAL TRIAL: NCT04671147
Title: Short-Term Preoperative Traction Method for Rigid and Severe Scoliosis: A Comparison Between Skull Tongs-Femoral Traction and Cotrel Longitudinal Traction
Brief Title: Short-Term Preoperative Traction Method for Rigid and Severe Scoliosis
Status: Completed | Type: Observational
Sponsor: Indonesian Orthopaedic Association (Other)
Responsible Party: Principal Investigator, Yoshi Pratama Djaja, Principal Investigator, Indonesian Orthopaedic Association
Other Study IDs: IndonesianOrthopaedic
Record Dates: First submitted 2020-11-28; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Scoliosis Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Skull tong femoral traction
  Interventions: Procedure: Preoperative traction
- Cotrell longitudinal traction
  Interventions: Procedure: Preoperative traction

INTERVENTIONS:
Procedure: Preoperative traction — Compare two methods of preoperative traction (Cotrel traction exercises and skull tongs femoral traction)

SUMMARY:
The investigators collected retrospective data of severe (>80o) and rigid scoliosis patients who underwent preoperative traction before correction surgery from 2016 to 2018. The first group consisted of patients who underwent Cotrel traction exercises and second group underwent continuous-progressively increasing Skull Tongs Femoral Traction (STFT) traction. Posterior fusion was performed in all patients. Intraoperative parameters (blood loss, operation time and level instrumented) and radiologic change (initial, post-traction and postoperative Cobb Angle) was evaluated and analyzed

ELIGIBILITY:
Inclusion Criteria:

* adolescence/adult idiopathic scoliosis;
* severe and rigid scoliosis (defined as Cobb angle more than 80° and flexibility index less than 25%);
* either skull tongs-femoral traction or Cotrel longitudinal traction used in the preoperative time period

Exclusion Criteria:

* other types of scoliosis (neuromuscular scoliosis, congenital scoliosis, etc.)
* intradural abnormalities (diastomatomyelia, tethered cord, etc)
* history of previous spine surgery

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: severe (>80o) and rigid scoliosis patients who underwent preoperative traction before correction surgery from 2016 to 2018
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Radiologic change | - Baseline - Immediately after 2 weeks of preoperative traction - immediately after the correction surgery
  Preoperative, post traction and postoperative xray

SECONDARY OUTCOMES:
Blood loss | Intraoperative
  The amount of blood loss during the correction surgery
Duration of surgery | Intraoperative
  The time required to perform the correction surgery
Number of instrumented levels | Intraoperative
  the number of vertebrae instrumented during the correction surgery